CLINICAL TRIAL: NCT05335590
Title: Adherence and Clinical Correlates in Persons With HIV on TAF
Acronym: ACT
Status: Active, not recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 22-0422
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Hiv
Keywords: HIV/AIDS; Adherence; TAF; Dried Blood Spots
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood in EDTA tube
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, 48-week, prospective study of PWH treated with TAF in which the investigators will compare TFV-DP concentrations in DBS in virologically suppressed vs. non-suppressed individuals and evaluate the utility of TFV-DP in DBS to predict future viremia. To accomplish this, the investigators will approach PWH currently taking TAF (which is being prescribed by a primary care physician) and who present to the clinic for regular HIV care and HIV VL assessment. Participants will complete up to 3 visits (at least 2 weeks apart) during the 48-week study follow-up period.

DETAILED DESCRIPTION:
Antiretroviral (ARV) drug exposure is directly linked to individual host factors, including age, weight, diet, and genetics. However, the main factor influencing long-term drug exposure is drug adherence. Adherence is a strong predictor of HIV treatment outcomes, but measuring adherence is difficult due to the inaccuracy of self-reporting and other commonly used monitoring methods. There is no gold-standard measure to monitor ARV exposure and adherence that has been implemented in clinical practice. Tenofovir diphosphate (TFV-DP), the phosphorylated anabolite of tenofovir (TFV), has distinct pharmacological characteristics that make it an ideal candidate for drug adherence and exposure monitoring. The long half-life of TFV-DP (~17 days) in red blood cells (RBC), which are abundant in dried blood spots (DBS) are properties that make it well suited for monitoring average TFV exposure over time both from tenofovir disoproxil fumarate (TDF) and tenofovir alafenamide (TAF). TFV-DP in DBS in persons with HIV (PWH) on TDF has been associated with viral suppression and is predictive of future viremia, even in patient who are virologically-suppressed. However, data on TFV-DP in DBS from TAF are lacking. To address this gap, this study will assess the association of TFV-DP in DBS from PWH on TAF with clinically-relevant virologic outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Females or males with HIV (≥18 years), able to give informed consent and comply with study procedures who are having a blood draw as part of their regular clinical care.
2. Being prescribed TAF-based ART >= 3 months.

Exclusion Criteria:

1. For females, active pregnancy or intent to become pregnant.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We propose a 48-week observational study at the University of Colorado Hospital Infectious Diseases Group Practice (UCH-IDGP) in PWH taking TAF. Its goals are to define the association between TFV-DP in DBS and viral suppression and future viremia.
Sampling Method: Non-Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Adjusted Odds Ratio of Level of Tenofovir-diphosphate (TFV-DP) in Dried Blood Spots (DBS) Associated with odds of HIV viral suppression at all study visits | 48 weeks
  HIV viral load, binary cutoff at assay level of detection (<20 copies/mL vs >= 20 copies/mL); reference group lowest adherence category for TFV-DP; adjusted odds ratio calculated using generalized estimated equations; concentration cutoffs established in prior research of healthy volunteers and persons with HIV (PWH)
Adjusted Odds Ratio of Level of Tenofovir-diphosphate (TFV-DP) in Dried Blood Spots (DBS) Associated with odds of HIV viremia at next study visit | 48 weeks
  HIV viral load, binary cutoff at assay level of detection (<20 copies/mL vs >= 20 copies/mL); reference group lowest adherence category for TFV-DP; adjusted odds ratio calculated using generalized estimated equations; concentration cutoffs established in prior research of healthy volunteers and persons with HIV (PWH)

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Anderson, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Health, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Coyle RP, Morrow M, Mann SC, Mainella V, Ellis SL, Schwab S, Coppinger C, Barker N, Ellison L, Zheng JH, Al Zuabi S, Alpert PE, Carnes TC, Buffkin DE Jr, Chai PR, Bushman LR, Kiser JJ, MaWhinney S, Brooks KM, Anderson PL, Castillo-Mancilla JR. Tenofovir-Diphosphate and Emtricitabine-Triphosphate Adherence Benchmarks in Dried Blood Spots for Persons With HIV Receiving Tenofovir Alafenamide and Emtricitabine-Based Antiretroviral Therapy (QUANTI-TAF). Clin Infect Dis. 2024 Nov 22;79(5):1233-1241. doi: 10.1093/cid/ciae212. PMID 38636950